CLINICAL TRIAL: NCT03256253
Title: An Open-Label Pilot Study of Pregabalin as Treatment for Alcohol Use Disorder
Brief Title: Pregabalin as Treatment for Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, John Mariani MD, Research psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7491
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol use disorder; alcohol abuse; treatment; lyrica
MeSH Terms: conditions — Alcoholism | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: open label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- pregabalin (Experimental): pregabalin up to daily dose of 600 mg
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — pregabalin up to 600 mg/day
  Other Names: lyrica

SUMMARY:
The proposed protocol is an 8 week open label outpatient pilot trial of the safety and efficacy of pregabalin (Lyrica) in the treatment of alcohol use disorder. The primary objective of the study is to determine the efficacy of pregabalin in promoting alcohol abstinence among individuals with an alcohol use disorder.

DETAILED DESCRIPTION:
The proposed protocol is an open label outpatient pilot trial of the safety and efficacy of pregabalin (Lyrica) in the treatment of alcohol use disorder. Pregabalin is commonly used for the treatment of pain issues such as fibromyalgia (chronic pain in your body), diabetic nerve pain, spinal cord injury nerve, and pain after shingles. We plan to enroll 20 participants in an 8-week trial.The ideal dosing, tolerability, and safety of pregabalin will be tested in outpatients with Alcohol Use Disorder (AUD). The primary objective of the study is to determine the efficacy of pregabalin in promoting alcohol abstinence among individuals with an alcohol use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-5 criteria for current alcohol use disorder
* Reports drinking a minimum of 5 standard drinks for men or 4 standard drinks for women at least 4 days per week over the past 28 days
* Between the ages of 18 and 65
* Able to provide informed consent and comply with study procedures

Exclusion Criteria:

* Subjects with any current psychiatric disorder as defined by DSM-5, other than AUD, that in the investigator's judgment might require intervention over the course of the study.
* Subjects receiving psychotropic medication treatment
* Evidence of moderate-to-severe alcohol withdrawal (CIWA-Ar > 13)
* History of alcohol withdrawal seizures or alcohol withdrawal delirium
* History of allergic reaction to candidate medication (pregabalin)
* Pregnancy, lactation, or failure in females patients to use adequate contraceptive methods
* Unstable physical disorders which might make participation hazardous
* Subjects who have a current DSM-5 diagnosis of moderate or severe substance use disorder, with the exception of alcohol, nicotine and caffeine use disorders. A diagnosis of a mild substance use disorder will not be exclusionary, as long as the current primary substance use disorder is alcohol.
* Are legally mandated to participate in alcohol use disorder treatment program
* Cognitively impaired

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: john mariani, md, Principal Investigator — new york psychiatric institute
Locations (1):
- Columbia Univeristy-STARS, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mariani JJ, Pavlicova M, Choi CJ, Brooks DJ, Mahony AL, Kosoff Z, Naqvi N, Brezing C, Luo SX, Levin FR. An open-label pilot study of pregabalin pharmacotherapy for alcohol use disorder. Am J Drug Alcohol Abuse. 2021 Jul 4;47(4):467-475. doi: 10.1080/00952990.2021.1901105. Epub 2021 Jun 5. PMID 34092158

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregabalin
Started | 18
Completed | 6
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 1
  Unknown or Not Reported | 4
Education [Mean (Standard Deviation); unit: years] | 14.1 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Dose of Pregabalin:
Description: Defined as the highest amount of medication per day maintained for a 7 day period.
Time Frame: over the course of the 8 week trial or participants' length of participation
Population: Data was available for 14 patients
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Pregabalin
Number analyzed (Participants) | 14
milligrams | 571.4 (80.2)

ADVERSE EVENTS:
Time Frame: Over the course of the 8 week trial or length of participant's participation
Description: Data was collected for 15 participants with post-enrollment data
Arm/Group | Pregabalin
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 12/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=15)
drowsiness (General disorders) | 4 (4)
fogginess (General disorders) | 3 (3)
dizziness (General disorders) | 3 (3)
insomnia (General disorders) | 3 (3)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
blurred vision (Eye disorders) | 2 (2)
vivid dreams (General disorders) | 2 (2)
dry mouth (General disorders) | 2 (2)
fatigue (General disorders) | 2 (2)
difficulty concentrating (General disorders) | 1 (1)
dry eyes (General disorders) | 1 (1)
eye infection (Eye disorders) | 1 (1)
increased sensitivity to alcohol (General disorders) | 1 (1)
swollen feet (General disorders) | 1 (1)
eye redness (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT03256253/SAP_000.pdf
  • Study Protocol (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT03256253/Prot_001.pdf